CLINICAL TRIAL: NCT00502216
Title: Naltrexone and Varenicline: Weight Gain and Tolerability in Smokers
Brief Title: Naltrexone and Varenicline: Weight Gain and Tolerability in Cigarette Smokers
Status: Completed | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: Yale University (Other)
Collaborators: National Institute on Alcohol Abuse and Alcoholism (NIAAA) (NIH); National Institute on Drug Abuse (NIDA) (NIH)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: 0704002538; P50AA015632 (NIH); NIH Grant P50-AA15632; NIH Grant K12-DA00167
Record Dates: First submitted 2007-07-13; First posted 2007-07-17 (Estimated); Results first posted 2010-09-21 (Estimated); Last update posted 2018-01-17 (Actual); Status verified 2018-01

CONDITIONS: Smoking; Nicotine Dependence
Keywords: Tobacco; Smoking; Weight; Naltrexone; Varenicline
MeSH Terms: conditions — Smoking; Tobacco Use Disorder; Body Weight | interventions — Naltrexone; Varenicline

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- 1 (Experimental): Arm 1 (Experimental) = Varenicline (Chantix) 1 mg oral tablet twice per day + naltrexone 25 mg oral capsule once per day
  Interventions: Drug: Naltrexone; Drug: Varenicline
- 2 (Placebo Comparator): Arm 2 (Placebo Comparator) = Varenicline (Chantix) 1 mg oral tablet twice per day + placebo naltrexone 25 mg oral capsule once per day
  Interventions: Drug: Varenicline

INTERVENTIONS:
Drug: Naltrexone — Varenicline (Chantix) 1 mg oral tablet twice per day + naltrexone 25 mg oral capsule once per day
  Arms: 1
Drug: Varenicline — Arm 1 (Experimental) = Varenicline (Chantix) 1 mg oral tablet twice per day + naltrexone 25 mg oral capsule once per day; Arm 2 (Placebo Comparator) = Varenicline (Chantix) 1 mg oral tablet twice per day + placebo naltrexone 25 mg oral capsule once per day
  Other Names: Chantix

SUMMARY:
The purpose of this study is to determine whether the combination of naltrexone (Depade) and varenicline (Chantix) minimizes post-smoking cessation weight gain and how well the combination is tolerated.

DETAILED DESCRIPTION:
Varenicline, a medication recently approved by the FDA, results in smoking cessation rates as high as 50%, significantly better than bupropion or placebo. However, varenicline does not reduce post-cessation weight gain, so weight concerns may keep some smokers from taking advantage of this effective therapy.

A potential solution would be to combine varenicline with an agent that reduces weight gain. In this regard, several studies have shown that naltrexone reduces weight gain (O'Malley et al., 2006; Toll et al., 2007).

This effect appears to be dose dependent, favoring lower doses (i.e., 25 mg daily). Thus, the proposed study seeks to conduct a pilot clinical trial of low dose naltrexone (25 mg daily) compared to placebo for minimizing weight gain in combination with varenicline for smoking cessation. Forty individuals who smoke at least 10 cigarettes per day will receive open-label varenicline for 12 weeks according to the recommended titration schedule up to 1 mg varenicline twice daily. Subjects will be randomized to receive either placebo or 25 mg naltrexone daily, with treatment starting at the quit date (after 1 week on varenicline to minimize nausea, a side effect of both varenicline and naltrexone) and continuing for 11 weeks. Subjects will take 12.5 mg naltrexone daily for the first week and 25 mg naltrexone daily for the next 10 weeks of treatment. In an effort to uncover mechanisms for naltrexone's weight suppressant effects, an experiment will be conducted using food odors and food consumption to examine naltrexone's effects on palatability, incentive value, and alliesthesia.

This experiment will be conducted pretreatment and after 2 weeks on naltrexone. The primary aim of this pilot study is to examine weight gain in participants who complete the clinical trial treatment. Weight gain for those who are continuously abstinent for the last 4 weeks of treatment and rates of adverse events will be secondary outcomes. The effects of naltrexone on odor/food palatability, incentive value, and alliesthesia will be exploratory outcomes. Effect size estimates for weight gain will be generated for a NIH grant application.

ELIGIBILITY:
Inclusion Criteria:

1. Between the ages of 18 and 75
2. Smoking 10 or more cigarettes per day
3. Fewer than 3 months of smoking abstinence in the past year
4. Motivated to stop smoking

Exclusion Criteria:

1. Current use of opiates, and/or a urine toxicology screen positive for opiates
2. Chronic pain conditions necessitating opioid treatment (naltrexone, an opioid antagonist will make these medications ineffective)
3. Evidence of significant hepatocellular injury as evidence by AST or ALT >3 x normal or elevated bilirubin
4. History of cirrhosis
5. Any serious or unstable disease within 6 months
6. Seizure risk
7. Diabetes mellitus requiring insulin or oral hypoglycemic medications
8. Hepatic or renal impairment
9. Use of a monoamine oxidase inhibitor in the prior 14 days
10. Clinically significant cardiovascular disease within 6 months
11. Uncontrolled hypertension
12. Baseline systolic blood pressure higher than 150 mm Hg or diastolic blood pressure higher than 95 mm Hg
13. Severe chronic obstructive pulmonary disease
14. History of cancer (except treated basal cell or squamous cell carcinoma of the skin)
15. History of clinically significant allergic reactions
16. Major depressive disorder within the past year requiring treatment
17. History of or current panic disorder, psychosis, bipolar disorder, or eating disorders
18. Alcohol or drug abuse/dependency within the past year
19. Use of another investigational drug within 30 days
20. Intention to donate blood or blood products during the treatment phase of the study
21. Use of tobacco products other than cigarettes or use of marijuana
22. Use of nicotine replacement therapy, clonidine, varenicline, bupropion, or nortriptyline within the month prior to enrollment or intention to use medication that might interfere with study medication
23. Body Mass Index (calculated as weight in kilograms divided by the square of height in meters) less than 15 or greater than 38 or weight less than 45 kg.
24. Females of childbearing potential who are pregnant, nursing, or not practicing effective contraception (oral injectable, or implantable contraceptives, intrauterine device, or barrier method with spermacide)

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 40 (Actual)
Dates: Start 2007-07; Primary Completion 2009-06 (Actual); Study Completion 2009-06 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Benjamin A. Toll, PhD, Principal Investigator — Yale University
Locations (1):
- Yale University School of Medicine Substance Abuse Treatment Unit, New Haven, Connecticut, United States

REFERENCES:
- [Derived] Livingstone-Banks J, Fanshawe TR, Thomas KH, Theodoulou A, Hajizadeh A, Hartman L, Lindson N. Nicotine receptor partial agonists for smoking cessation. Cochrane Database Syst Rev. 2023 May 5;5(5):CD006103. doi: 10.1002/14651858.CD006103.pub8. PMID 37142273

RESULTS

PARTICIPANT FLOW:
Groups:
- Varenicline + Naltrexone: Arm 1 (Experimental) = Varenicline (Chantix) 1 mg oral tablet twice per day + naltrexone 25 mg oral capsule once per day
- Varenicline + Placebo: Arm 2 (Placebo Comparator) = Varenicline (Chantix) 1 mg oral tablet twice per day + placebo naltrexone 25 mg oral capsule once per day
Period: Overall Study
Arm/Group | Varenicline + Naltrexone | Varenicline + Placebo
Started | 21 | 19
Completed | 21 | 19
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Varenicline + Naltrexone | Varenicline + Placebo | Total
Number analyzed (Participants) | 21 | 19 | 40
Age, Continuous [Mean (Standard Deviation); unit: years] | 50.29 (11.08) | 42.42 (9.57) | 46.55 (11.00)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 15 | 12 | 27
  Male | 6 | 7 | 13
Region of Enrollment [Number; unit: participants]
  United States | 21 | 19 | 40

OUTCOME MEASURES:

1. Primary Outcome: Weight Gain in Treatment Completers
Time Frame: baseline and 12 weeks
Population: Subpopulation of participants who reported quitting smoking
Measure: Mean (Standard Deviation); unit: Pounds
Arm/Group | Varenicline + Naltrexone | Varenicline + Placebo
Number analyzed (Participants) | 17 | 11
Pounds | 3.35 (6.61) | 4.14 (5.15)

2. Secondary Outcome: Weight Gain in Participants Who Are Continuously Abstinent for the Last 4 Weeks of Treatment
Time Frame: 4 weeks
Population: Analyzed are those that remained abstinent for last 4 weeks of treatment
Measure: Mean (Standard Deviation); unit: pounds
Arm/Group | Varenicline + Naltrexone | Varenicline + Placebo
Number analyzed (Participants) | 3 | 3
pounds | 0 (4.36) | 7.67 (2.31)

3. Secondary Outcome: Tolerability of the Combination of 25 mg Naltrexone and 2 mg Varenicline
Description: Tolerability was measured by tracking adverse events. These data are reported in detail in the adverse events section. Presented are an unduplicated count of participants that experienced at least 1 adverse event.
Time Frame: 11 weeks
Measure: Count of Participants; unit: Participants
Arm/Group | Varenicline + Naltrexone | Varenicline + Placebo
Number analyzed (Participants) | 21 | 19
Participants | 10 | 4

ADVERSE EVENTS:
Arm/Group | Varenicline + Naltrexone | Varenicline + Placebo
Serious Adverse Events (participants affected / at risk) | 0/21 | 0/19
Other Adverse Events (participants affected / at risk) | 10/21 | 4/19
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk, or affected / at risk where a term's number at risk differs:
Term (organ system) | Varenicline + Naltrexone (N=21) | Varenicline + Placebo (N=19)
Nausea (General disorders) | 6 | 0/0
Anxiety (Psychiatric disorders) | 3 | 1
Constipation (Gastrointestinal disorders) | 3 | 1
Fatigue (General disorders) | 4 | 0
Depression (Psychiatric disorders) | 3 | 0
Flatulence (Gastrointestinal disorders) | 2 | 1
Insomnia (Psychiatric disorders) | 3 | 0
Joint pain (General disorders) | 2 | 1
Sleepiness (Psychiatric disorders) | 2 | 0
Vivid dreams (Psychiatric disorders) | 2 | 0
Acid reflux (Gastrointestinal disorders) | 0 | 1
Other (General disorders) | 2 | 1
Decreased Appetite (Metabolism and nutrition disorders) | 1 | 0
Dizzyness (Nervous system disorders) | 1 | 0
Drowsiness (General disorders) | 1 | 0
Dry Mouth (General disorders) | 1 | 0
Headache (General disorders) | 1 | 0
Increased Appetite (Metabolism and nutrition disorders) | 1 | 0
Nightmares (General disorders) | 1 | 0
Sweating (General disorders) | 1 | 0
Vomiting (Gastrointestinal disorders) | 1 | 0

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes; Agreement restricts PI disclosure of results: No